CLINICAL TRIAL: NCT00972569
Title: Specific Aims 3: Define in Hospitalized Decompensated CHF Patients With Renal Dysfunction, the Renal Actions of Low Dose Intravenous Infusion of BNP in the Presence and Absence of Acute PDE V Inhibition in Improving Renal Function
Brief Title: Low Dose Intravenous (IV) Infusion of BNP in the Presence and Absence of Acute Type V Phosphodiesterase (PDE V) in Improving Renal Function in Hospitalized Chronic Heart Failure (CHF) Patients With Renal Dysfunction
Acronym: Aim 3 BNP/PDEV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Horng Chen, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-003303; 1R01HL08415501A2
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure; Renal Dysfunction
Keywords: BNP with or without PDE-V in heart failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Natriuretic Peptide, Brain; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BNP with PDE-V (Active Comparator): BNP (Nesiritide) will be infused starting at 0.0025 g/Kg/min IV for 3 hours, if tolerated increased to 0.005 g/kg/min for 45 hours without bolus with PDEV inhibition, they will also receive Sildenafil 12.5 mg at timepoints 0,12, 24 and 36 hours
  Interventions: Drug: BNP and PDE-V
- BNP (Nesiritide) will be infused at 0.005 u/Kg/min IV for 48 h (Active Comparator): BNP (Nesiritide) will be infused at 0.025 ug/Kg/min IV for 3 hours then 0.005ug/kg/min 45 hours without bolus. No PDE-V is given.
  Interventions: Drug: BNP
- standard care (No Intervention): Patients randomized to this group will continue to receive therapy at the discretion of the heart failure specialist who is managing the patient (with the exception of BNP and low dose dopamine). Blood and Urine will be collected after the patient has been randomized for 48 hours

INTERVENTIONS:
Drug: BNP and PDE-V — low dose BNP 0.025 u/kg/min for 3 hours then 0.005ug/kg/min 45 hours PDE-V 12.5 mg 4 time points
  Other Names: nesiritide (Natrecor); Viagra
  Arms: BNP with PDE-V
Drug: BNP — low dose BNP at 0.025 u/kg/min if tolerated then at 0.005 ug/kg/min for 45 hours
  Other Names: Nesiritide (Natrecor)
  Arms: BNP (Nesiritide) will be infused at 0.005 u/Kg/min IV for 48 h

SUMMARY:
The purpose of the study is to determine if low doses of BNP can improve renal function in people with chronic heart failure with renal dysfunction, also to determine whether Sildenafil assists with improvement. This study will enroll only hospitalized patients with heart failure.

DETAILED DESCRIPTION:
The broad objective of this protocol is to advance our understanding of the pathophysiological mechanisms of human Cardiorenal Syndrome (CRS) with a specific emphasis upon the biological interaction between diuretic therapy, the renin-angiotensin-aldosterone-system (RAAS) and cyclic 3'-5'-guanosine monophosphate (cGMP) pathway.

Chronic heart failure (CHF) as a result of left ventricular systolic dysfunction is a clinical syndrome with high mortality and morbidity. Renal dysfunction is a common and progressive complication of CHF and despite growing recognition of the frequent presentation of combined cardiac and renal dysfunction, or "Cardiorenal Syndrome (CRS)", its underlying pathophysiology is not well understood, with a lack of consensus as to its appropriate management.

The main objective of this study is to extend the findings of the applicant's studies in both human and experimental CHF and determine if low dose intravenous (IV) (0.005/Kg/min) administration of BNP in hospitalized decompensated CHF patients with renal dysfunction would improve the renal function. Furthermore, based on our preliminary data, we also sought to assess if PDE V inhibition potentiated these renal enhancing actions.

Hypothesis: Low dose IV infusion of BNP in hospitalized decompensated CHF patients with CRS will enhance renal and humoral functions as compared to standard therapy, which will be further potentiated by PDEV inhibition as evident by:

Increased sodium excretion, Increased creatinine clearance Decreased plasma creatinine and blood urea nitrogen Suppression of the renin-angiotensin-aldosterone system, Increased renal cGMP generation

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to St Mary's Hospital, Mayo Clinic Rochester MN with NYHA class III-IV decompensated CHF with renal dysfunction as Calculated creatinine clearance of equal or less than 60 ml/min but greater than 20 ml/min using the Cockcroft-Gault formula.

Exclusion Criteria:

* Cause of acute renal dysfunction can be reasonably ascribed to factors other than heart failure or its treatment
* Known intrinsic renal diseases or renal artery stenosis of =>50%
* Patients taking Nitrates within the previous 24 hours
* Patients needing emergency coronary revascularization or those who may have rapidly changing cardiac function (i.e. patients with acute myocardial infarction or shock)
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Systolic blood pressure < 90 mmHg or cardiogenic shock.
* Requirement of pressors for maintenance of blood pressure.
* Intra-aortic blood pump use.
* History of significant uncorrected renal artery stenosis as defined by >50% stenosis.
* Severe aortic or mitral stenosis or significant LV outflow tract obstruction. Hgb < 10 mg/dL
* Pregnant or nursing women.
* Contraindication to nesiritide.
* Inability to have NSAID dose held for up to 30 hours, if being treated with these medications.
* Administration of radiocontrast medium within 7 days of enrollment or anticipated use of such agents during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this aim will be a comparison of the 3 groups for the percent change in creatinine clearance, and blood urea nitrogen from baseline to 48 hours. | each blood and urine collections 4 time points

SECONDARY OUTCOMES:
The secondary endpoints for this aim will be a comparison of the 3 groups for the percent change in plasma, sodium excretion, aldosterone, and renal cGMP generation from baseline line to 48 hours | each blood and urine collection at 4 time points

CONTACTS AND LOCATIONS:
Overall Officials: Dr Horng H Chen, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- [Derived] Hubers SA, Benike SL, Johnson BK, McKie PM, Scott C, Chen HH. Renal Effects of Combination Phosphodiesterase V Inhibition and Low-Dose B-Type Natriuretic Peptide in Acute Heart Failure: A Randomized Clinical Trial. Circ Heart Fail. 2024 Dec;17(12):e011761. doi: 10.1161/CIRCHEARTFAILURE.124.011761. Epub 2024 Nov 8. PMID 39513267
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials